CLINICAL TRIAL: NCT04673565
Title: A Randomized Controlled Trial Evaluating the Effects of Motivational Interviewing in New Hearing Aid Users
Brief Title: Motivational Interviewing in Hearing Aid Users
Acronym: MI-HAT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Desmond A Nunez, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H20-02393
Record Dates: First submitted 2020-12-13; First posted 2020-12-17 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Hearing Loss; Motivation; Hearing Disability; Hearing Disorders and Deafness
MeSH Terms: conditions — Hearing Loss; Hearing Disorders; Deafness | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant
Masking Description: The study will be a multi-center, prospective, randomized patient-blind controlled trial and employ a between-subject, pretest-posttest design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Control groups that undergo standard audiological care
- Treatment (Experimental): Treatment groups that undergo motivational interviewing with audiological care
  Interventions: Behavioral: Motivational interviewing

INTERVENTIONS:
Behavioral: Motivational interviewing — Each participant in the treatment group will attend a 1-hour MI group session with 9 other participants hosted by a practicing MI therapies via Zoom at one month after the initial visit. This session will utilize MI to elicit motivation in each participant. Participants will also receive standard care delivered at in-person audiology clinic visits.
  Arms: Treatment

SUMMARY:
Hearing loss is one of the most common chronic disabilities in the older adult population and affects their quality of life. Hearing aid use can improve one's quality of life by increasing a person's ability to detect, differentiate and locate sound, and improve speech recognition. Several factors seem to reduce motivation to use a hearing aid. Fears of exclusion and shame due to hearing loss are major deterrents to hearing aid use. Motivational interviewing (MI) is a counselling style aimed at creating desire in patients to change their behavior.

There have been pilot studies that suggest one-on-one MI can increase hearing aid use, but other pilot studies found the reverse hence the evidence is inconclusive. The effectiveness of group MI therapy is also being investigated in MI research. While results in group MI research are promising, studies investigating group MI have been limited to substance abuse.

DETAILED DESCRIPTION:
Hearing loss is one of the most common chronic disabilities in the older adult population and affects their quality of life. Hearing aid use can improve one's quality of life by increasing a person's ability to detect, differentiate and locate sound, and improve speech recognition. Several factors seem to reduce motivation to use a hearing aid. Fears of exclusion and shame due to hearing loss are major deterrents to hearing aid use. MI is a counselling style aimed at creating desire in the patient to change their behavior.

To our knowledge, there have been no studies that investigated the impact of group MI on hearing aid use.

Hypothesis Standard care with motivational interviewing in a group setting does not alter the hearing aid usage when compared to the standard care alone in the new hearing aid users.

Study Methodology

Trial Objectives:

The purpose of this study is to determine the efficacy of group MI in improving adherence to hearing aid use, and to report the adverse effects of group MI if they exist.

Trial Design

1. Settings The study will be a multi-center, prospective, randomized patient-blind controlled trial and employ a between-subject, pretest-posttest design.

   Study participants will be recruited at the audiology clinics located within the greater Vancouver region, BC. Audiology clinics will comply with Work safe BC and the Provincial Health Officer's COVID-19 orders as related to safety plans and best practices.
2. Sample size determination Previous pilot research by Aazh (2016) suggests using a conservative estimation of effect size where d = 0.6 to estimate the sample size. A sample size of 180 participants (n = 90 in each group) will be required to achieve a level of significance of p = 0.05, power of 90%, at a randomization ratio of 1:1 and allowing for a 50% drop-out rate. We use a higher dropout rate than Aazh's study (50% vs. 20%) to compensate for the uncertainty surrounding COVID-19 pandemic. The estimated period for recruitment, intervention and data acquisition for this study is 48 months.
3. Outcomes Differences in hearing aid use hours will be measured at each time point. This is a quantitative measure indicated by the mean number of hours the aid is used as recorded by the hearing aids' data logging feature. For bilateral hearing aid users, the mean number of hours will be calculated by averaging the left and right hearing aid use hours.

   Participants will also be asked to fill out the International Outcome Inventory for Hearing Aids (IOI-HA) questionnaire (Cox & Alexander, 2002) at each time point. This self-reported questionnaire is designed to measure the effectiveness of hearing aid interventions. The IOI-HA have been rigorously tested for their validity, reliability, and sensitivity (Cox & Alexander, 2002; Vestergaard, 2006).
4. Randomization Individuals who meet the inclusion criteria and provide informed consent will be assigned to a non-identifiable number sequence. Each sequence will have been previously allocated using block randomization to either treatment or control groups using a statistical software package, such as STATA. Block size variation will be used to prevent prediction of treatment. Creation of allocation lists will be done by the study coordinator, who will not be involved in data collection.

   * Treatment Group (MI group session + Standard care) Each participant in the treatment group will attend a 1-hour MI group session with 9 other participants hosted by a practicing MI therapies via Zoom at one month after the initial visit. This session will utilize MI to elicit motivation in each participant. Participants will also receive standard care delivered at in-person audiology clinic visits.
   * Control Group (Standard care) Each participant in the control group will receive standard care as typically delivered by audiologists at in-person audiology clinic visits. No additional treatment will be provided.
5. Statistical Analysis Descriptive Statistics (means, standard deviation, frequency) will be used to summarize sample statistics. Repeated Measures (RM)-ANOVA tests will be conducted at each sampling interval to determine if there is a significant difference between the intervention and control groups with respect to the average number of hours the hearing aids are activated per day. Pearson's correlations will also be used to measure the strength of associations between hearing aid use hours via the data-logging feature and self-reported measures via the IOI-HA questionnaire. Data will be analyzed using STATA.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* New hearing aid user
* Unilateral or bilateral hearing threshold above 25 dB in the worse ear (based on four-frequency PTA across 0.5, 1, 2 and 4 kHz, high-frequency PTA across 3, 4, 6, and 8 kHz, and low-frequency PTA across 0.5, 1 and 2 kHz)

Exclusion Criteria:

* History of hearing aid use
* Do not understand the English language
* Unable to complete the online questionnaires in English language
* Have inconsistent pure-tone audiometric readings
* Have medical constraints that prohibit them from wearing hearing aids

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-03-16 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Hearing aid use hours | Study assessments will be performed during the initial visit, and at 1, 3, 6 and 12-month time points.
  Differences in hearing aid use hours will be measured at each time point
Patient reported outcomes | Study assessments will be performed during the initial visit, and at 1, 3, 6 and 12-month time points.
  International Outcome Inventory for Hearing Aids questionnaire (Cox & Alexander, 2002) at each time point.

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aazh H. Feasibility of conducting a randomized controlled trial to evaluate the effect of motivational interviewing on hearing-aid use. Int J Audiol. 2016;55(3):149-56. doi: 10.3109/14992027.2015.1074733. Epub 2015 Sep 2. PMID 26328620
- [Background] Cox RM, Alexander GC. The International Outcome Inventory for Hearing Aids (IOI-HA): psychometric properties of the English version. Int J Audiol. 2002 Jan;41(1):30-5. doi: 10.3109/14992020209101309. PMID 12467367
- [Background] Vestergaard MD. Self-report outcome in new hearing-aid users: Longitudinal trends and relationships between subjective measures of benefit and satisfaction. Int J Audiol. 2006 Jul;45(7):382-92. doi: 10.1080/14992020600690977. PMID 16938796
- [Derived] Liu AQ, Wijesinghe P, Lee M, Lau C, Sun J, Nunez DA. A randomized controlled trial evaluating the effects of motivational interviewing in new hearing aid users (MI-HAT): study protocol for a randomized controlled trial. Trials. 2023 May 22;24(1):346. doi: 10.1186/s13063-023-07352-7. PMID 37217960